CLINICAL TRIAL: NCT03030183
Title: A Phase 2 Multicenter, Open-Label, Uncontrolled Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of RA101495 in Subjects With Paroxysmal Nocturnal Hemoglobinuria Who Have an Inadequate Response to Eculizumab
Brief Title: Phase 2 Safety and Efficacy Study of Zilucoplan (RA101495) to Treat PNH Patients Who Have an Inadequate Response to Eculizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA101495-01.203
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zilucoplan (RA101495) (Experimental): Subjects will receive RA101495 at the dose of 0.3 mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC
  Interventions: Drug: Zilucoplan (RA101495)

INTERVENTIONS:
Drug: Zilucoplan (RA101495) — 0.3 mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of RA101495 in patients with paroxysmal nocturnal hemoglobinuria (PNH) who have an inadequate response to eculizumab. Patients will be treated with RA101495 for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PNH by flow cytometry
* Inadequate response to eculizumab defined as having received eculizumab for at least 6 months plus a documented LDH level ≥ 1.5 x the upper limit of normal (ULN) and/or the presence of a known C5 mutation conferring resistance to eculizumab

Exclusion Criteria:

* History of meningococcal disease
* Current systemic infection or suspicion of active bacterial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anita Hill, Study Chair — St James' Institute of Oncology
Locations (6):
- United States (6):
  - Investigative Site, Duarte, California
  - Investigative Site, Los Angeles, California
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Manhasset, New York
  - Investigative Site, Durham, North Carolina
  - Investigative Site, Dallas, Texas

REFERENCES:
- See also: Related Info — https://learningcenter.ehaweb.org/eha/2018/stockholm/214782/anita.hill.ra101495.a.subcutaneously-administered.peptide.inhibitor.of.html?f=menu=14*media=3*speaker=664274

RESULTS

PARTICIPANT FLOW:
Groups:
- Zilucoplan (RA101495): Subjects will receive zilucoplan (RA101495) at the dose of 0.3 mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC
  Zilucoplan (RA101495): 0. 3mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC
Period: Overall Study
Arm/Group | Zilucoplan (RA101495)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Zilucoplan (RA101495): Subjects will receive zilucoplan (RA101495) at the dose of 0.3 mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC
  Zilucoplan (RA101495): 0.3 mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC
Arm/Group | Zilucoplan (RA101495)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
Weight [Mean (Standard Deviation); unit: kg] | 109.67 (13.97)
Height [Mean (Standard Deviation); unit: cm] | 176.20 (7.60)
BMI [Mean (Standard Deviation); unit: kg/m2] | 35.72 (7.76)

OUTCOME MEASURES:

1. Primary Outcome: Change-from-baseline in Serum Lactate Dehydrogenase (LDH) Levels.
Description: Change-from-baseline through Week 12 in serum lactate dehydrogenase (LDH) levels
Time Frame: Through Week 12 of the study
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Zilucoplan (RA101495)
Number analyzed (Participants) | 3
U/L | 100.3 (128.0)

2. Secondary Outcome: Change-from-baseline Bilirubin Values
Description: Changes from baseline at each of the scheduled postbaseline time-points
Time Frame: Through week 12
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Zilucoplan (RA101495)
Number analyzed (Participants) | 3
umol/L
  Week 1 | -3.3 (5.1)
  Week 2 | -4.7 (12.0)
  Week 3 | -4.3 (7.5)
  Week 4 | -0.3 (2.9)
  Week 6 | -6.7 (17.5)
  Week 8 | -2.3 (12.5)
  Week 10 | -7.7 (14.8)
  Week 12 | -2.0 (6.2)

3. Secondary Outcome: Change-from-baseline Total Hemoglobin Values
Description: Changes from baseline at each of the scheduled postbaseline time-points
Time Frame: Through week 12
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Zilucoplan (RA101495)
Number analyzed (Participants) | 3
g/L
  Week 1 | 5.7 (4.2)
  Week 2 | 3.3 (3.8)
  Week 3 | 0.3 (4.0)
  Week 4 | -0.3 (7.2)
  Week 6 | 0.7 (5.8)
  Week 8 | -3.3 (4.2)
  Week 10 | 2.3 (3.1)
  Week 12 | 0.3 (2.5)

4. Secondary Outcome: Change-from-baseline Free Hemoglobin Values
Description: Changes from baseline at each of the scheduled postbaseline time-points
Time Frame: Through week 12
Population: Efficacy Evaluable
Measure: Number; unit: mg/dL
Arm/Group | Zilucoplan (RA101495)
Number analyzed (Participants) | 3
mg/dL
  Week 1: number analyzed (Participants) | 1
  Week 1 | -145.90
  Week 2: number analyzed (Participants) | 1
  Week 2 | -140.60
  Week 3: number analyzed (Participants) | 1
  Week 3 | -147.70
  Week 4: number analyzed (Participants) | 1
  Week 4 | -138.40
  Week 6: number analyzed (Participants) | 1
  Week 6 | -147.30
  Week 8: number analyzed (Participants) | 1
  Week 8 | -148.10
  Week 10: number analyzed (Participants) | 1
  Week 10 | -143.50
  Week 12: number analyzed (Participants) | 1
  Week 12 | -144.30

5. Secondary Outcome: Change-from-baseline Haptoglobin Values
Description: Changes from baseline at each of the scheduled postbaseline time-points
Time Frame: Through week 12
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Zilucoplan (RA101495)
Number analyzed (Participants) | 3
g/L
  Week 1 | 0.000 (0.000)
  Week 2 | 0.000 (0.000)
  Week 3 | 0.000 (0.000)
  Week 4 | 0.133 (0.231)
  Week 6 | 0.000 (0.000)
  Week 8 | 0.000 (0.000)
  Week 10 | 0.000 (0.000)
  Week 12 | 0.000 (0.000)

6. Secondary Outcome: Change-from-baseline Reticulocyte Values
Description: Changes from baseline at each of the scheduled postbaseline time-points
Time Frame: Through week 12
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Zilucoplan (RA101495)
Number analyzed (Participants) | 3
10^12 cells/L
  Week 1 | -0.0190 (0.0382)
  Week 2 | 0.0090 (0.0052)
  Week 3 | 0.0430 (0.0327)
  Week 4 | 0.0477 (0.0499)
  Week 6 | 0.0310 (0.0157)
  Week 8 | 0.0253 (0.0248)
  Week 10 | 0.0350 (0.0350)
  Week 12 | 0.0190 (0.0092)

7. Secondary Outcome: Change-from-baseline Hemoglobinuria Values
Description: Changes from baseline at each of the scheduled postbaseline time-points Hemoglobinuria was assessed using a urine colorimetric scoring system with a score of 1 through 10. Where 1 represents no hemoglobinuria and 10 represents maximum hemoglobinuria.
Time Frame: Through week 12
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zilucoplan (RA101495)
Number analyzed (Participants) | 3
score on a scale
  Week 1: number analyzed (Participants) | 1
  Week 1 | 0.0
  Week 2: number analyzed (Participants) | 2
  Week 2 | 0.5 (0.7)
  Week 3: number analyzed (Participants) | 2
  Week 3 | 0.5 (0.7)
  Week 4: number analyzed (Participants) | 2
  Week 4 | 1.0 (1.4)
  Week 6: number analyzed (Participants) | 2
  Week 6 | 0.5 (0.7)
  Week 8: number analyzed (Participants) | 1
  Week 8 | 2.0
  Week 10 | 2.3 (2.5)
  Week 12 | -0.3 (2.1)

ADVERSE EVENTS:
Time Frame: Through week 12 of the Study
Arm/Group | Zilucoplan (RA101495)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilucoplan (RA101495) (N=3)
Nausea (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Haemoglobinuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's right to discuss or publish trial results after the trial is completed. Disclosure agreements are negotiated separately with each PI

DOCUMENTS (2):
  • Study Protocol (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT03030183/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03030183/SAP_001.pdf